CLINICAL TRIAL: NCT00910481
Title: Balloon Pump Assisted Coronary Intervention Study
Acronym: BCIS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Cardiovascular Intervention Society (Other)
Responsible Party: Principal Investigator, Dr Divaka Perera, Professor of Cardiology, British Cardiovascular Intervention Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN40553718; ISRCTN40553718
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Left Ventricular Dysfunction
Keywords: Coronary Artery Disease; Percutaneous Transluminal Coronary Angioplasty; Intraaortic Balloon Pumping; Left Ventricular Dysfunction; High Risk
MeSH Terms: conditions — Coronary Artery Disease; Ventricular Dysfunction, Left | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Elective IABP Insertion (Experimental)
  Interventions: Device: Intra-Aortic Balloon Pump
- No Planned IABP Insertion (No Intervention)

INTERVENTIONS:
Device: Intra-Aortic Balloon Pump — Elective IABP insertion before PCI
  Arms: Elective IABP Insertion

SUMMARY:
This study will test the hypothesis that elective use of the Intra-Aortic Balloon Pump (IABP) in patients undergoing high-risk Percutaneous Coronary Intervention (PCI) will reduce the rate of in-hospital major adverse cardiac and cerebrovascular events compared to patients who are managed without planned insertion of IABP.

ELIGIBILITY:
Inclusion Criteria:

* impaired left ventricular function (Ejection Fraction < 30%)
* large area of myocardium at risk (BCIS-1 Myocardial Jeopardy Score ≥ 8/12)

Exclusion Criteria:

* cardiogenic shock
* acute STEMI within previous 48 hours
* complications of recent AMI (including ventricular septal defect, severe mitral regurgitation, intractable ventricular arrhythmias)
* contraindications to IABP use (including significant iliac or femoral arterial disease and more than mild aortic regurgitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2005-12; Primary Completion 2011-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Divaka Perera, MRCP, MD, Principal Investigator — Guy's and St Thomas' Hospital NHSFT, London, UK; Simon Redwood, FRCP, MD, Principal Investigator — Guy's and St Thomas' Hospital NHSFT, London, UK; Rodney Stables, FRCP, DM, Principal Investigator — Liverpool Cardiothoracic Centre, Liverpool, UK; Martyn Thomas, FRCP, MD, Principal Investigator — Guy's and St Thomas' Hospital NHSFT, London, UK
Locations (1):
- British Cardiovascular Intervention Society, London, United Kingdom

REFERENCES:
- [Result] Perera D, Stables R, Clayton T, De Silva K, Lumley M, Clack L, Thomas M, Redwood S; BCIS-1 Investigators. Long-term mortality data from the balloon pump-assisted coronary intervention study (BCIS-1): a randomized, controlled trial of elective balloon counterpulsation during high-risk percutaneous coronary intervention. Circulation. 2013 Jan 15;127(2):207-12. doi: 10.1161/CIRCULATIONAHA.112.132209. Epub 2012 Dec 6. PMID 23224207
- [Result] Perera D, Stables R, Thomas M, Booth J, Pitt M, Blackman D, de Belder A, Redwood S; BCIS-1 Investigators. Elective intra-aortic balloon counterpulsation during high-risk percutaneous coronary intervention: a randomized controlled trial. JAMA. 2010 Aug 25;304(8):867-74. doi: 10.1001/jama.2010.1190. PMID 20736470
- [Derived] Perera D, Stables R, Booth J, Thomas M, Redwood S; BCIS-1 Investigators. The balloon pump-assisted coronary intervention study (BCIS-1): rationale and design. Am Heart J. 2009 Dec;158(6):910-916.e2. doi: 10.1016/j.ahj.2009.09.015. PMID 19958856

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elective IABP Insertion | No Planned IABP Insertion
Started | 151 | 150
Completed | 151 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Elective IABP Insertion: Left ventricular ejection fraction was 23.6% (SD, 5.2%) in the elective IABP group
- No Planned IABP Insertion: Left ventricular ejection fraction was 23.6% (SD, 5.5%) in the no planned IABP group
- Total: Total of all reporting groups
Arm/Group | Elective IABP Insertion | No Planned IABP Insertion | Total
Number analyzed (Participants) | 151 | 150 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 33 | 59
  >=65 years | 125 | 117 | 242
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 122 | 117 | 239

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac and Cerebrovascular Events
Description: (composite endpoint of death, acute myocardial infarction, further revascularization or cerebrovascular event)
Time Frame: Hospital discharge or 28 days following PCI, whichever occurs sooner
Population: All
Measure: Count of Participants; unit: Participants
Arm/Group | Elective IABP Insertion | No Planned IABP Insertion
Number analyzed (Participants) | 151 | 150
Participants | 23 | 24

2. Secondary Outcome: All-cause Mortality
Time Frame: 6-months following randomization
Reporting Status: Not Posted

3. Secondary Outcome: Major Procedural Complications
Time Frame: Duration of PCI procedure
Reporting Status: Not Posted

4. Secondary Outcome: Bleeding Complications (Major and Minor)
Time Frame: Hospital Discharge or 28 days following PCI (whichever occurs sooner)
Reporting Status: Not Posted

5. Secondary Outcome: Access Site Complications
Time Frame: Hospital Discharge or 28 days following PCI (whichever occurs sooner)
Reporting Status: Not Posted

6. Secondary Outcome: Transient Ischemic Attack
Time Frame: Hospital Discharge or 28 days following PCI (whichever occurs sooner)
Reporting Status: Not Posted

7. Secondary Outcome: Length of Hospital Stay
Time Frame: Hospital Discharge
Reporting Status: Not Posted

8. Secondary Outcome: Procedural Success
Time Frame: Duration of PCI procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Elective IABP Insertion | No Planned IABP Insertion
All-Cause Mortality (participants affected / at risk) | 3/151 | 1/150
Serious Adverse Events (participants affected / at risk) | 2/151 | 0/150
Other Adverse Events (participants affected / at risk) | 2/151 | 16/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elective IABP Insertion (N=151) | No Planned IABP Insertion (N=150)
CVA (Nervous system disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elective IABP Insertion (N=151) | No Planned IABP Insertion (N=150)
Procedural Complications (Cardiac disorders) | 2 | 16 — Overall, rescue IABP insertion was required in 18 patients assigned to have no planned IABP insertion, including 13 for procedural hypotension, 1 for pulmonary edema, and 1 for sudden vessel closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No